CLINICAL TRIAL: NCT02587377
Title: New Biomarkers for Invasive Fungal Infections in Paediatric Haemato-oncology. A National Belgian Study
Brief Title: New Biomarkers for Invasive Fungal Infections in Paediatric Haemato-oncology
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The current rate of recruitment is insufficient.
Sponsor: Queen Fabiola Children's University Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HU14
Record Dates: First submitted 2014-06-03; First posted 2015-10-27 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2014-09

CONDITIONS: Haemato-oncological Paediatric Patients Under Intensive Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort 1 (Other): single cohort of patient
  Interventions: Other: Non Standard of Care blood samples collection

INTERVENTIONS:
Other: Non Standard of Care blood samples collection — According to Belgian Law of 07MAY2004, if non standard of care interventions are performed as per protocol, the study must be classified as Interventional Study.

SUMMARY:
The availability of sensitive and specific fungal biomarkers could be a precious help to improve the management of patients suffering from fungal diseases, not only by allowing preemptive treatment, but also by offering objective elements to assess patient therapeutic response and prognosis.

The use of such biomarkers could also contribute to accurately evaluate novel antifungal drugs effectiveness and to serve as a valuable tool to guide decisions regarding ineffective treatments and dose selection in product development. Using two or three tests may increase the sensitivity to detect IFI.

The results of the serum assays will be correlated to the definition of 'proven' fungal infection as defined by the EORTC/MSG criteria published in 2008. Based upon results from adults' studies, the investigators estimate that galactomannan antigen or 1, 3 β-D glucan could reasonably have a 90% sensitivity (with a 95% CI between 73% and 98%) under the current design. As concern the aspergillus fumigatus PCR, sensitivity and specificity could be estimated between 63% to 100% and 87% to 96.7%, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Any febrile episode in :

   * either a neutropenic child suffering from acute lymphoblastic leukemia under induction chemotherapy or relapse, acute myeloblastic leukemia under chemotherapy (all cycles of chemotherapy included) or myelodysplasic syndrome
   * an allogenetic hematopoietic stem cell transplantation recipient child, from conditioning till 3 months or receiving aggressive immunosuppressive therapy for at least 1 months
2. Age of children will be from 3 months till 18 years
3. Informed consent from the parents and from children older than 12 years obtained

Exclusion Criteria:

1. Any previous history of fungal infection (proven, probable or possible) with prescription of secondary oral prophylaxis (voriconazole or posaconazole) under current use at the time of the study.
2. Any previous episode already enrolled (only one episode/patient).

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2013-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
clinical relevance of a "combined tests strategy" (positive results of serum 1,3 beta-D-glucan test and/or PCR Aspergillus fumigatus, with or without positive galactomannan antigen) to improve early diagnosis of IFI | 1 year after the end of the study
  To assess the clinical relevance, in term of sensitivity and specificity, of a "combined tests strategy" (positive results of serum 1,3 beta-D-glucan test and/or PCR Aspergillus fumigatus, with or without positive galactomannan antigen) to improve early diagnosis of IFI and to allow a pre-emptive "diagnostic driven" therapeutic approach among haemato-oncological immunocompromised children.

SECONDARY OUTCOMES:
% of early diagnosis of invasive fungal infection using serum 1,3 beta-D-glucan test | 1 year after the end of the study
Validity of the PCR for A. fumigatus in early diagnosis of invasive aspergillosis in a pediatric population. | 1 year after the end of the study
incidence of invasive fungal infection among neutropenic febrile episodes reported | 1 year after the end of the study